CLINICAL TRIAL: NCT01246973
Title: Oral Curcumin for Radiation Dermatitis in Breast Cancer Patients
Brief Title: Oral Curcumin for Radiation Dermatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Julie Ryan, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: URCC 10054; URCC 09005 (Other: NCI); U10CA037420 (NIH); URCC 10054 (Other: University of Rochester); NCT01238198 (obsolete NCT alias)
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Radiation-induced Dermatitis
Keywords: Oral Curcumin; Radiation Dermatitis; Breast Cancer Patients
MeSH Terms: conditions — Radiodermatitis | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- curcumin (Experimental): 4 Curcumin C3 Complex 500mg capsules (2.0 g) taken orally 3 times/day throughout course of radiation treatments plus one week
  Interventions: Drug: Curcumin
- Placebo (Placebo Comparator): 4 placebo capsules taken orally 3 times/day throughout course of radiation treatments plus one week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Curcumin — 4 Curcumin C3 Complex 500mg capsules (2.0 g) taken orally 3 times/day throughout course of radiation treatments plus one week
  Other Names: Curcumin C3 Complex
  Arms: curcumin
Drug: Placebo — 4 placebo capsules taken orally 3 times/day throughout course of radiation treatments plus one week
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether curcumin, an ingredient of some foods, can prevent or reduce the severity of skin reactions (dermatitis) caused by radiation therapy. Dermatitis is a common side effect of radiation treatment, but few effective treatments have been developed for it. Curcumin is a natural compound found in both turmeric and curry powder. It has been used for centuries as a spice (curry), a food coloring and as a food preservative. Curcumin is non-toxic and has been found to enhance the functions of normal tissues..

DETAILED DESCRIPTION:
Radiation is a toxic agent and a widely accepted form of treatment for various types of cancer. Approximately half of all women with breast cancer receive radiation therapy. Despite advances in medical technology, radiation therapy still causes severe skin effects. Radiation dermatitis occurs in approximately 90% of patients and ranges in severity from mild redness to more severe skin changes. Dermatitis is a common side effect of radiation treatment, but few effective treatments have been developed for it; currently, there is no standard treatment for the prevention of radiation-induced dermatitis. Curcumin is a natural compound found in both turmeric and curry powder. It has been used for centuries as a spice (curry), a food coloring and as a food preservative. Curcumin is non-toxic and has been found to enhance the functions of normal tissues.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of non-inflammatory breast adenocarcinoma (including in situ and bilateral)
* scheduled to begin radiotherapy without concurrent chemotherapy; concurrent hormone or Herceptin® (trastuzumab)treatment is okay
* can have been treated by lumpectomy or mastectomy with or without adjuvant or neoadjuvant chemotherapy or hormonal treatment
* can have had breast reconstruction
* scheduled to receive 25-35 radiation treatment sessions (1 session per day) using standard irradiation fractionation (1.8-2.0 Gy per sessions) OR 16-20 radiation treatment sessions (1 session per day) using Canadian irradiation fractionation (2.2-3.0 Gy per session)(100, 101).
* able to swallow medication.
* three weeks must have elapsed after chemotherapy and surgery before the patient can begin the study
* able to understand English

Exclusion Criteria:

* inflammatory breast cancer
* previous radiation therapy to the breast or chest
* concurrent chemotherapy treatment
* concurrent treatment with anti-coagulants (e.g., coumadin®, warfarin®), or anti-EGFR (human epidermal growth factor receptor) drugs (e.g. Iressa® (gefitinib), Erbitux® (cetuximab, C225); aspirin is allowed
* known radiosensitivity syndromes (e.g., Ataxia-telangiectasia)
* collagen vascular disease, unhealed surgical sites, or breast infections

Ages: 21 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Actual)
Dates: Start 2011-02; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Ryan, PhD, MPH, Principal Investigator — University of Rochester

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Curcumin | Placebo
Started | 344 | 342
Completed | 283 | 295
Not Completed | 61 | 47
Not completed — Other | 38 | 25
Not completed — Adverse Event | 16 | 9
Not completed — Withdrawal by Subject | 7 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Curcumin | Placebo | Total
Number analyzed (Participants) | 344 | 342 | 686
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (0.6) | 57.7 (0.5) | 57.6 (0.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 344 | 342 | 686
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 264 | 237 | 501
  Unknown or Not Reported | 74 | 98 | 172
Race/Ethnicity, Customized [Number; unit: participants]
  White/caucasian | 307 | 293 | 600
  black/african american | 29 | 30 | 59
  other race | 8 | 19 | 27
Region of Enrollment [Number; unit: participants]
  United States | 344 | 342 | 686

OUTCOME MEASURES:

1. Primary Outcome: Mean Radiation Dermatitis Severity Score
Description: The outcome measures will be the severity of radiation dermatitis, using the Radiation Dermatitis Score (RDS), at the end of treatment in each treatment arm. (Objective: To examine the efficacy of curcumin in preventing and/or reducing the severity of dermatitis in radiation treatment site in breast cancer patients). The RDS score ranges from 0-4 with higher scores indicating worse outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 283 | 295
units on a scale | 2.02 (0.05) | 1.99 (0.06)
Statistical Analysis 1: Comparison: Curcumin vs Placebo; Test type: Superiority or Other; p = 0.6555, F-test

2. Secondary Outcome: Percentage of Subjects With Moist Desquamation
Description: Moist desquamation was measured by the presence of wet, patchy crusting, oozing, or ulcerated skin in areas where skin was peeling in sheets.
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 283 | 295
percentage of participants | 9.541 | 12.203
Statistical Analysis 1: Comparison: Curcumin vs Placebo; Test type: Superiority or Other; p = 0.3504, Chi-squared

ADVERSE EVENTS:
Arm/Group | Curcumin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/344 | 0/342
Other Adverse Events (participants affected / at risk) | 0/344 | 0/342

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes